CLINICAL TRIAL: NCT05631483
Title: A Feasibility Study for the DAISe Thrombectomy Device in Colombia
Brief Title: COlombia DAISe FEasibility Exercise
Acronym: COFEE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment/Recruitment
Sponsor: MIVI Neuroscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101929
Record Dates: First submitted 2022-10-19; First posted 2022-11-30 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Stroke, Acute Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DAISe (Experimental): DAISe Thrombectomy Device
  Interventions: Device: DAISe

INTERVENTIONS:
Device: DAISe — Use of the DAISe Thrombectomy Device

SUMMARY:
This study is to assess initial safety and performance data of the DAISe Thrombectomy Device for removal of thrombus during an acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Pre-stroke (24 hours prior to stroke onset) independent functional status in activities of daily living with modified Rankin Score 0-2.
* Diagnosis of acute ischemic stroke with study enrollment time < 8 hours from onset of symptoms.
* Disabling stroke defined as a baseline NIHSS > 6.
* Confirmed symptomatic, large vessel occlusion of the intracranial internal carotid artery, middle cerebral artery, M1.
* Signed informed consent from patient or legal representative.

Exclusion Criteria:

* Computed tomography (CT) or Magnetic Resonance Imaging (MRI) evidence of recent/ fresh hemorrhage on presentation.
* Clinical history, past imaging or clinical judgment suggests that the intracranial occlusion is chronic.
* Rapidly improving neurological deficits based on the investigator's clinical judgement.
* Pregnancy; if a woman is of child-bearing potential and urine or serum beta HCG test is positive.
* Severe contrast allergy or absolute contraindication to iodinated contrast.
* Difficult endovascular access, difficult aortic arch or severe neurovascular tortuosity that will result in an inability to deliver endovascular therapy.
* Evidence of dissection in the carotid or target artery for treatment.
* Presence of a carotid artery stenosis or occlusion requiring balloon angioplasty or stenting at time of the procedure.
* Renal failure (serum creatinine level ≥ 3 mg/dL or on dialysis).
* Severe, sustained hypertension resistant to treatment (SBP >185 mmHg or DBP>110 mmHg).
* Use of warfarin anticoagulation with International Normalized Ratio (INR) >3.0 at the time of the procedure or any known hemorrhagic or coagulation deficiency.
* Use of a direct thrombin inhibitor within the last 48 hours; partial thromboplastin time (PTT) > 2.0 times the normal prior to procedure.
* Cerebral vasculitis or evidence of active systemic infection.
* Suspicion of aortic dissection, presumed septic embolus or suspicion of bacterial endocarditis.
* Clinical symptoms suggestive of bilateral stroke or occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation).
* A severe or fatal comorbid illness that will prevent improvement or follow-up or that will render the procedure unlikely to benefit the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Rate of Successful Revascularization | Procedure
  mTICI (Modified TICI) 2b-3 of the target vessel post-treatment with the DAISe Thrombectomy Device
Rate of Symptomatic Intracranial Hemorrhage | 24 hours post-procedure

SECONDARY OUTCOMES:
Rate of Procedure related Complications | Through 90 day post-procedure
Occurrence of all intracranial hemorrhage | 24 hours post-procedure
All-cause mortality | Through Acute Hospital Discharge
Embolization to a New Vascular Territory | Procedure
Successful Revascularization after first attempt with DAISe | Procedure
  mTICI (modified TICI) 2b-3 after first pass with device
Successful Revascularization after first attempt with DAISe | Procedure
  mTICI (modified TICI) 2c-3 after first pass with device
Successful Revascularization at end of procedure | Procedure
  mTICI (modified TICI) 2b-3 at the end of procedure
Successful Revascularization at end of procedure | Procedure
  mTICI (modified TICI) 2c-3 at the end of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Boris Pabon, MD, Principal Investigator — Angiosur
Locations (1):
- Angiosur - Unidad Vascular Integral, Itagüí, Antioquia, Colombia